CLINICAL TRIAL: NCT07018440
Title: The Effect of Low Volume Oral Carbohydrate Feeding on Nausea, Vomiting and Recovery in Bariatric Surgery Patients: A Randomized Controlled Trial
Brief Title: Low-Volume Oral Carbohydrate Feeding in Bariatric Surgery: Effects on PONV and Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OrCarBariatricNBSN
Record Dates: First submitted 2025-05-23; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Bariatric Surgery; Postoperative Nausea and Vomiting
Keywords: Perioperative Nursing; Bariatric Surgery; Postoperative Nausea and Vomiting; Postoperative Recovery; Carbohydrate Feeding
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: This study used a randomized, parallel-group design with two arms: an intervention group receiving low-volume oral carbohydrate loading before surgery, and a control group receiving standard care. Participants were allocated using computer-generated block randomization, and each participant received only one type of intervention.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, no blinding was applied to participants or investigators. However, outcome assessors and statisticians were blinded to group allocation to reduce bias during data analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Carbohydrate Feeding Group (Experimental): Oral administration of 200 ml 12.5% carbohydrate solution 2 hours before surgery.
  Interventions: Dietary Supplement: Low-Volume Oral Carbohydrate Loading (200 mL of 12.5% solution)
- Control Group (No Intervention): No carbohydrate solution provided; only standard fasting and care applied.

INTERVENTIONS:
Dietary Supplement: Low-Volume Oral Carbohydrate Loading (200 mL of 12.5% solution) — Patients were given Low Volume Oral Carbohydrate feeding (200 mL 12.5% solution) in the preoperative period.
  Arms: Carbohydrate Feeding Group

SUMMARY:
This randomized controlled trial aims to evaluate the effects of preoperative oral administration of 200 ml 12.5% carbohydrate solution on postoperative nausea, vomiting, and recovery in bariatric surgery patients. The intervention group received carbohydrate loading two hours before surgery. Outcomes were measured using the Rhodes Index of Nausea, Vomiting and Retching (RINVR) and the Postoperative Recovery Index (PORI).

DETAILED DESCRIPTION:
This randomized controlled trial was designed to evaluate the effects of preoperative low-volume oral carbohydrate loading on postoperative nausea, vomiting, and recovery in patients undergoing bariatric surgery. A total of 105 adult patients scheduled for bariatric surgery were randomized into two groups: an intervention group (n = 53) and a control group (n = 52). The intervention group received 200 mL of a 12.5% carbohydrate solution orally two hours before surgery, while the control group followed standard preoperative fasting protocols without receiving any carbohydrate supplementation.

The primary hypothesis was that preoperative low-volume carbohydrate loading would reduce the frequency and severity of postoperative nausea, vomiting, and retching (PONV), and improve postoperative recovery. Data were collected using validated instruments including the Rhodes Index of Nausea, Vomiting and Retching (RINVR) and the Postoperative Recovery Index (PORI). Outcomes were assessed within 24 hours postoperatively and at postoperative day 30.

Randomization was performed using computer-generated block randomization, and outcome assessment was blinded. The intervention was administered by a trained researcher, and standard postoperative nursing care protocols were applied to both groups.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Scheduled for bariatric surgery
* ASA score ≤ IV
* Literate in Turkish and able to provide informed consent

Exclusion Criteria:

* Use of antiemetics, steroids, or opioids within 24 hours pre-op
* Need for ICU post-op
* Reoperation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
RINVR Total Score | Day 1
  RINVR Total Score within 24 hours postoperative
PORI Score | Day 30
  PORI Score at discharge and at 30-day follow-up

CONTACTS AND LOCATIONS:
Overall Officials: HAMDİYE BANU KATRAN, Principal Investigator — Marmara University
Locations (1):
- Istanbul Education and Research Hospital, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to confidentiality concerns and institutional policy.